CLINICAL TRIAL: NCT00542568
Title: Safety and Efficacy of Sustained Erythropoietin Therapy of Anemia in Chronic Kidney Disease Patients Using EPODURE Biopump
Brief Title: Safety and Efficacy of Sustained Erythropoietin Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medgenics Medical Israel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MG-001-02
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Cohort 1 (Low Dose group) 18-25 IU/kg/day
  Interventions: Biological: EPODURE (dermal Biopump for erythropoietin)
- 2 (Experimental): Cohort 2 (Intermediate Dose group): 35-45 IU/kg/day
  Interventions: Biological: EPODURE (dermal Biopump for erythropoietin)
- 3 (Experimental): Cohort 3 (High Dose group): 55-65 IU/kg/day
  Interventions: Biological: EPODURE (dermal Biopump for erythropoietin)

INTERVENTIONS:
Biological: EPODURE (dermal Biopump for erythropoietin) — Subjects will undergo similar study procedures and evaluations; however each dosage group will receive a different targeted dose of EPO delivered via EPODURE Biopump

SUMMARY:
The purposes of this study are to assess safety, efficacy, and subject satisfaction of EPODURE Biopump (an autologous dermal biopump capable of sustained secretion of therapeutic EPO in the body, using a small tissue explant from the patient's own skin) treatment in Chronic Kidney Disease (CKD) patients over a period of up to six (6) months.

DETAILED DESCRIPTION:
Anemia, is a common complication of chronic kidney disease (CKD) resulting from insufficient production of the hormone erythropoietin by the damaged kidney leading to a decrease in red blood cells production by the bone marrow.

Replacement therapy with recombinant human erythropoietin can effectively correct anemia in patients. However, despite the availability of recombinant human erythropoietin for more than a decade for use in CKD patients, two thirds of patients initiating dialysis have a hematocrit less than 30%, and three fourths have a hemoglobin (Hb) less than 11 g/dL the level recommended by the National Kidney Foundation Kidney Disease Outcome Quality Initiative. Treatment with recombinant human erythropoietin typically involves subcutaneous (SC) administration at regular intervals followed by frequent laboratory tests to monitor hemoglobin concentration. There is a need to provide an significantly improved care in this area using a sustained therapy approach.

EPODURE, is an autologous dermal biopump capable of sustained secretion of therapeutic EPO in the body, using a small tissue explant from the patient's own skin. The EPODURE biopump is harvested directly from the patient's dermis under local anesthetic. EPODURE Biopumps, produced by ex vivo transduction of MOs with Helper Dependent Adenoviral EPO vectors (HDAd-EPO), expresses and secretes EPO. The EPODURE Biopump is subsequently implanted subcutaneously back to the patient in order to provide continuous delivery of a known amount of EPO.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female subjects between 18 to 75 years of age at the time of screening visit.
2. Subject with Anemia of Chronic Renal Failure CKD stage 3-4. estimated GFR of 15-60 ml/min with Female: Hb < 10 g%, Male: Hb < 11 g%.
3. Chronic renal failure subjects who are EPO naïve or have been off EPO or similar Erythropoietic drugs for more than four (4) weeks.
4. Subjects who are clinically stable.
5. Adequate iron stores (transferrin saturation ≥ 20.0% and ferritin ≥100 ng/ml).
6. Subjects who receive anti-coagulation treatment may be enrolled provided anti-coagulation treatment can be discontinued two weeks prior to the harvesting visit. INR level must be within normal range (0.9 - 1.5).

Signed written informed consent to participate in the study by subject

Exclusion Criteria:

1. Uncontrolled hypertension (defined as diastolic blood pressure > 110 mmHg or systolic blood pressure > 180 mmHg during screening).
2. Congestive heart failure (New York Heart Association functional class III or IV).
3. Grand mal seizures within 2 years of the screening visit.
4. Clinical evidence of severe hyperparathyroidism as defined by PTH levels of > 10 times the upper normal limits.
5. Major surgery within 12 weeks of the screening visit.
6. Systemic hematologic diseases (e.g., sickle cell anemia, myelodysplastic syndromes, hematologic malignancy, myeloma, hemolytic anemia).
7. Current systemic infection, active inflammatory disease, or malignancy under treatment.
8. Known positivity for HIV antibody.
9. Subjects known to have tested positive at any time in the past for antibodies to erythropoietic proteins.
10. Subject has history of malignancy within the past 2 years prior to the screening visit, with the exception of basal cell carcinoma.
11. Subjects with other concurrent severe and/or uncontrolled medical condition which could compromise participation in the study (i.e. active infection, uncontrolled diabetes, uncontrolled hypertension, congestive cardiac failure, unstable angina, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months, uncompensated cirrhosis, active upper GI tract ulceration).
12. Subject is currently enrolled in, or has not yet completed a period of at least 30 days since ending other investigational device or drug trial(s).
13. Psychiatric, addictive, or any other disorder that compromises ability to give truly informed consent for participation in this study.
14. Female subjects of child-bearing potential and not having undergone permanent sterilization procedures.
15. Pregnant and lactating female subjects.
16. Chronic alcoholic or drug abuse subjects.
17. Steroid or other immunosuppressive treatment.
18. Subjects unwilling or unable to comply with the study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-08; Primary Completion 2012-07 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Safety Endpoints: adverse events; safety laboratory values; immune response by determination of anti-EPO antibodies; dermal safety outcomes | 6 weeks and 6 months

SECONDARY OUTCOMES:
Elevation of serum EPO levels at least 10 mU/ml above baseline for duration of at least six (6) weeks following implantation | 6 weeks and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Eithan Galun, M.D, Principal Investigator — Hadassah Medical Organization; Doron Schwartz, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (2):
- Israel (2):
  - Hadassah Medical Organization, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv